CLINICAL TRIAL: NCT05456425
Title: Multicenter, Double-Masked, Randomized, Vehicle-Controlled 12-Month Parallel Comparison of the Safety and Efficacy of 0.1% and 0.2% CBT-001 Versus Vehicle, Dosed Twice-Daily, in Patients With Pterygium
Brief Title: A Clinical Trial on Safety and Efficacy of CBT-001 in Patients With Pterygium
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cloudbreak Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBT-CS301
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Intervention Model Description: Multicenter, Double-Masked, Randomized, Vehicle-Controlled Parallel Comparison with dosing twice-daily in eye(s) with pterygium
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vehicle (Placebo Comparator): Emulsion eye drop without drug
  Interventions: Drug: Vehicle
- CBT-001 Low Dose (Experimental): CBT-001 eye drop
  Interventions: Drug: CBT-001
- CBT-001 High Dose (Experimental): CBT-001 eye drop
  Interventions: Drug: CBT-001

INTERVENTIONS:
Drug: CBT-001 — CBT-001 eye drop
  Arms: CBT-001 High Dose; CBT-001 Low Dose
Drug: Vehicle — Formulation without drug
  Arms: Vehicle

SUMMARY:
The objective is to evaluate the safety and efficacy of low dose and high dose CBT-001 eye drop dosed twice daily for 24 months compared to vehicle in reducing conjunctival hyperemia and preventing pterygium progression in eyes with pterygia.

DETAILED DESCRIPTION:
Clinical Hypotheses:

1. CBT-001 dosed twice daily is more effective than vehicle in:

   * Reducing conjunctival hyperemia by demonstrating a statistically significant difference and clinically relevant improvement in the mean severity grade change from baseline.
   * Preventing pterygium progression, by demonstrating a statistically significant and clinically relevant improvement on drug vs vehicle mean difference in the change in pterygium length from baseline.
2. CBT-001 dosed twice daily maintains the above efficacies and has an acceptable ocular and systemic safety and tolerability profile when administered topically.

ELIGIBILITY:
Inclusion Criteria:

Pterygium with conjunctival hyperemia

Exclusion Criteria:

Pterygium removal within the last 6 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
conjunctival hyperemia | 3 month
  Mean difference of conjunctival hyperemia grade change from baseline.
pterygium length | 12 month
  Mean difference of pterygium lesion length change from baseline.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (20):
  - Trinity Research Group, Dothan, Alabama
  - Horizon Eye Specialists & LASIK Center, Sun City, Arizona
  - West Coast Eye Institute, Bakersfield, California
  - Global Research Mangement, Glendale, California
  - Inland Eye Specialists, Hemet, California
  - Eye Research Foundation, Newport Beach, California
  - Shultz Chang Vision, Northridge, California
  - North Bay Eye Associates INC, Petaluma, California
  - Santa Barbara Eye Care, Santa Barbara, California
  - Advanced Research; LLC, Deerfield Beach, Florida
  - Bruce A. Segal, MD, Delray Beach, Florida
  - International Research Center, Tampa, Florida
  - The Eye Care Institute, Louisville, Kentucky
  - Center for Sight, Henderson, Nevada
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas
  - DCT-Shah Research, LLC dba Discovery Clinical Trials, McAllen, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - R and R Eye Research, San Antonio, Texas
  - Emerson Clinical Research Institute, LLC, Falls Church, Virginia
- Australia (5):
  - The Centre for Eye Research Australia, East Melbourne, Melbourne
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Bendigo Eye Clinic, Bendigo, Victoria
  - Sunshine Eye Surgeons, St Albans, Victoria
- China (10):
  - Beijing Tongren Hospital; CMU, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Hainan Provincial Eye Hospital, Haikou
  - 1st Affiliated Hospital of University of South China, Hengyang
  - The Second People's Hospital of Yunnan Province, Kunming
  - The First Affiliated Hospital of NC University, Nanchang
  - Eye Hospital of Shandong First Medical University, Qingdao
  - Eye Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College, Wuhan
  - Xiamen Eye Center of Xiamen University, Xiamen
- India (6):
  - Advanced Eye Centre PGIMER, Chandigarh, Chandigarh
  - Netralaya Super Specialty Eye Hospital, Ahmedabad, Gujarat
  - Narayana Nethralaya, Bangalore, Karnataka
  - L V Prasad Eye Institute, Bhubaneswar, Odisha
  - SP Medical College and AG of Hospitals, Bikaner, Rajasthan
  - Icare Eye Hospital, Noida, Uttar Pradesh
- New Zealand (3):
  - Auckland Eye, Auckland
  - Eye Institute, Auckland
  - Southern Eye Specialists, Christchurch

IPD SHARING:
Plan to Share IPD: No